CLINICAL TRIAL: NCT05166395
Title: Treatment of Surgical Scar With 2940 nm Erbium: Yttrium Aluminum Garnet (YAG) Laser Examined Under Optical Coherence Tomography
Brief Title: Laser Treated Scars and Optical Coherence Tomography (OCT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: device not available to initiate study.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Keyvan Nouri, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190751
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Scar
Keywords: surgical scar
MeSH Terms: conditions — Cicatrix | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Er:YAG laser Group (Experimental): The study is a split-scar model. Participants will have half of their lesion receive a total of three sessions using 2940 nm Er:YAG laser spaced over a 4-week study participation interval.
  Interventions: Device: Er:YAG laser
- Control (No Intervention) Group (No Intervention): The study is a split-scar model. Participants will serve as their own control and have half of their lesion receive no intervention.

INTERVENTIONS:
Device: Er:YAG laser — 2940 nm Er:YAG laser treatment spread over 3 sessions within 4 weeks on participant's scar on either the head/neck, trunk or extremities.
  Arms: Er:YAG laser Group

SUMMARY:
The purpose of this research study is to learn about the effects of the 2940 nm Erbium: Yttrium-Aluminum-Garnet (Er:YAG) laser on treating surgical scar using optical coherence tomography, a medical imaging device.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 years or older
2. Patients should have Fitzpatrick skin types of I-IV
3. Patients should have mild to severe post-surgical scarring located on head and neck
4. Scar lengths of at least 3 cm.
5. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. The patient should not be receiving any additional systemic, topical, or intralesional treatment of the scars during the study
2. Scar size less than 3 cm in length
3. Pregnant or lactating females
4. Fitzpatrick skin type of V-VI
5. Scleroderma
6. Photosensitivity
7. Botulinum toxin injection, facial laser resurfacing, chemical peels, fillers, or usage of oral retinoid within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
POSAS Scar Assessment | Up to 13 weeks
  Patient and Observer Scar Assessment Scale (POSAS) has a total score ranging from 6 (normal skin) to 60 (severely scarred skin).
Surgical Scar Blood Flow | Up to 13 weeks
  As measured using optical coherence tomography
Surgical Scar Skin Roughness | Up to 13 weeks
  As measured using optical coherence tomography
Surgical Scar Collagen Content | Up to 13 weeks
  As measured using optical coherence tomography
Surgical Scar Epidermal Thickness | Up to 13 weeks
  As measured using optical coherence tomography

SECONDARY OUTCOMES:
Incidence of Adverse Events | Up to 13 weeks
  Adverse events reported by participant and evaluated by treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Nouri, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No